CLINICAL TRIAL: NCT00506844
Title: A Phase II Study of Pre-Operative Concurrent Chemoradiotherapy With Cetuximab, Irinotecan, and Capecitabine in Resectable Rectal Cancer
Brief Title: Preoperative Chemoradiotherapy With Cetuximab in Rectal Cancer
Acronym: ERBIRIX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-165
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Rectal Neoplasms; Neoadjuvant Treatment
Keywords: Rectal neoplasms; Neoadjuvant treatment; Cetuximab; Irinotecan; Capecitabine; Radiotherapy; Combination chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Cetuximab; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab, Irinotecan, Capecitabine

SUMMARY:
This study is to estimate the pathologic complete response rate of cetuximab, irinotecan, and capecitabine concurrent with radiotherapy given preoperatively in patients with resectable rectal cancer.

DETAILED DESCRIPTION:
Daily fractions of radiotherapy at 1.8 Gy to total of 45 Gy to tumor and draining lymph nodes and followed by a coned-down boost of 5.4 Gy to the tumor are delivered concurrently with chemotherapy.

Cetuximab 400 mg/m2 is given intravenously on D-6 (1 week before radiation), followed by 250 mg/m2 once a week (D 1, 8, 15, 22 & 29).

Administration of irinotecan and capecitabine starts on day 1 of radiotherapy. Capecitabine is administered orally at a dose of 825 mg/m2 twice daily during weekdays (Monday to Friday) during radiotherapy. Irinotecan 40 mg/m2 is given intravenously once a week (D 1, 8, 15, 22 & 29).

Four to eight weeks after completion of chemoradiotherapy, curative surgery is performed.

Safety evaluation of the study will be performed after the first 6 patients treated. If more than 1 out of 6 patients received less than 70-80% of planned dose of capecitabine or irinotecan, the dosage of chemotherapy in the further study patients will be adjusted by a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum
* Distal margin of tumor located from 0 to 8 cm from anal verge
* Stage T3/T4 ± N+ by MRI ± endorectal ultrasonography
* ECOG performance status 0-2
* No prior chemotherapy, radiotherapy to pelvis, immunotherapy, and EGFR pathway targeting therapy
* Adequate organ functions
* Patients must sign the informed consent

Exclusion Criteria:

* Malignant disease of the rectum other than adenocarcinoma or arisen from chronic inflammatory bowel disease
* Any defined hereditary colorectal cancer
* Any unresected synchronous colon cancer
* R0 resection of tumor is not clinically possible
* Any distant metastasis
* Intestinal obstruction or impending obstruction, but decompressing colostomy is permitted
* Any previous or concurrent malignancy other than non-melanoma skin cancer or in situ cancer of uterine cervix
* Any other morbidity or situation with contraindication for chemoradiotherapy
* Patients with history of significant gastric or small bowel resection, or malabsorption syndrome, or other lack of integrity of the upper gastrointestinal tract that may compromise the absorption of capecitabine
* History of severe pulmonary disease
* Pregnant or lactating women or patients of childbearing potential not predicting adequate contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05; Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Pathologic stage Tumor regression grade | After operation

SECONDARY OUTCOMES:
Toxicity measured by NCICTC v3 | During chemoradiation
Disease-free survival | Three year

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hae Jung, M.D.Ph.D, Principal Investigator
Locations (4):
- South Korea (4):
  - National Cancer Center Korea, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul